CLINICAL TRIAL: NCT03828890
Title: A Pilot Study to Assess Screening for Diabetic Retinopathy Using Retinal Camera in Family Medicine Clinic
Brief Title: Assess Screening for Diabetic Retinopathy Using Retinal Camera in Family Medicine Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bryan Farford, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-009449
Record Dates: First submitted 2019-01-16; First posted 2019-02-04 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Trial (Other): Intervention includes screening eye exam using Optos technology
  Interventions: Other: Screening eye exam using Optos technology

INTERVENTIONS:
Other: Screening eye exam using Optos technology — Retinal imaging using Optos technology to identify Diabetic Retinopathy

SUMMARY:
The long-term goal for this study is to improve compliance of screening for diabetic retinopathy among subjects with diabetes. Researchers are also doing this research to determine the ability of appropriately trained family physicians to screen for and identify Diabetic Retinopathy using a retinal camera in addition to determining an overall patient perspective of the convenience and cost-effectiveness of retinal imaging within a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age
* Diabetes Mellitus Type I or II
* Patient is willing and able to provide informed written consent

Exclusion Criteria:

• Known Diabetic Retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Family Physicians Screening for Diabetic Retinopathy - Number of photographs that are interpreted accurately by the family physicians when compared to the retinal specialist | 6 months.
  Number of photographs that are interpreted accurately by the family physicians when compared to the retinal specialist. These photographs are obtained using retinal imaging and after the initial read by the family physicians trained to interpret the images, the images will be reviewed by the retinal specialist to determine if the interpreted results are accurate.

SECONDARY OUTCOMES:
Screening Impact - Percentage increase in the screening rates for Diabetic Retinopathy using retinal imaging. | 6 months
  Percentage increase in the screening rates for Diabetic Retinopathy using retinal imaging using OPTOS when compared with the traditional dilated eye exam.The current screening rate is around 55%.

OTHER OUTCOMES:
Patient Satisfaction | 6 months
  Percentage change in patient satisfaction and how much are patients willing to pay out of pocket to screen for Diabetic Retinopathy using retinal imaging. Each patient will be surveyed and these questions will help determine patient satisfaction and their willingness to pay for this versus usual care. We will ask the following questions:
  1. Did you find the Retinal Imaging an easy/efficient way of screening for eye disease as a result of having diabetes? Yes/No
  2. If you had to pay for this out-of-pocket what is the maximum amount you would be willing to pay?
     1. $25
     2. $50
     3. $75
     4. $100
     5. >$100 This will help us determine the patient's level of satisfaction and their willingness to pay out of pocket for the service.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Farford, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials